CLINICAL TRIAL: NCT04780854
Title: Drug Repurposing for the Prevention of Chemotherapy-induced Peripheral Neuropathy (CIPN)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Collaborators: German University in Cairo (Other)
Responsible Party: Principal Investigator, Sara Araby Ramadan Aly Mosa, Bsc., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: S-5-2020
Record Dates: First submitted 2020-11-02; First posted 2021-03-04 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: Cancer; chemotherapy-induced peripheral neuropathy; metformin; neuropathy
MeSH Terms: conditions — Neoplasms | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Metformin group (Active Comparator): 1 gm metformin tablet administered twice daily for 3 months
  Interventions: Drug: Metformin
- Metformin-free (Placebo Comparator): 1 placebo tablet administered twice daily for 3 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Participants in the intervention group will be administered metformin tablets 2 gm daily during the chemotherapy treatment duration
  Other Names: N,N-dimethylbiguanide; Cidophage
  Arms: Metformin group
Drug: Placebo — Participants in the placebo group will be administered metformin free tablet as placebo twice daily
  Other Names: inactive pill
  Arms: Metformin-free

SUMMARY:
Chemotherapy cause many adverse events including induction of peripheral neuropathy. Metformin, the AMPK activator, was found to have protective effect against chemotherapy induced peripheral neuropathy in mouse model and in clinical trials as well. There are different hypothesized mechanisms through which metformin does the protective effect. Such as enhancing mitochondrial activity, reduction of ROS and nitric oxide and activation of AMPK.

DETAILED DESCRIPTION:
Chemotherapy can cause a variety of side effects. One of the most common side effects is Chemotherapy induced peripheral neuropathy (CIPN), it commonly caused by Paclitaxel chemotherapy which is usually used in the treatment of breast cancer. Metformin which is known as a safe anti-diabetic drug, was found to have a protective effect on neurons. It gave positive results in chemotherapy induced peripheral neuropathy in mouse models and in some clinical trials

ELIGIBILITY:
Inclusion Criteria:

* Age (18-75) male and female patients
* Scheduled to be treated with single agent Paclitaxel
* Performance status according to Eastern Cooperative oncology group (ECOG) < 2.
* Patients who are willing and able to review and provide written consent, patients who can read the questionnaires

Exclusion Criteria:

* Previous exposure to chemotherapy drugs that cause neuropathy, patients treated with medications that increase the risk of neuropathy like amiodarone, Colchicine, metronidazole, phenytoin.
* Patients with impaired liver functions or kidney functions.
* Patients with a history of any serious adverse events or interaction or hypersensitivity to Metformin.
* Pregnant or lactating females.
* Patients who are using metformin for any other cause.
* Patients with sensory or motor neuropathy of any grade prior to enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2020-11-03 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of grade 2-4 neurotoxicity in both arms | 3 months
  Measured by NCI-CTCAE system

SECONDARY OUTCOMES:
Difference in biological markers in both arms. | 3 months
  Measurement of Nerve growth factor (NGF)
Difference in biological markers in both arms. | 3 months
  Measurement of Malondialdehyde (MDA)
Percentage of Qulaity of Life (QOL) deterioration in both arms | 3 months
  Measured using Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - Neurotoxicity (FACT/GOG-NTX) questionnaire. The higher the score, the better the quality of life.
Percentage of other treatment related common adverse events in both arms. | 3 months
  Graded using NCI-CTCAE system

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed H. Solayman, PhD. Pharm., Study Chair — German University in Cairo; Loay M. Kassem, PhD, Principal Investigator — Cairo University; Danira Ashraf Habashy, PhD Pharm., Principal Investigator — German University in Cairo; Sara A. Mosa, Bsc, Principal Investigator — German University in Cairo
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaballah A, Shafik A, Elhusseiny K, Ashraf M. Chemotherapy-Induced Peripheral Neuropathy in Egyptian Patients: Single Institution Retrospective Analysis. Asian Pac J Cancer Prev. 2018 Aug 24;19(8):2223-2227. doi: 10.22034/APJCP.2018.19.8.2223. PMID 30139229
- [Background] Mao-Ying QL, Kavelaars A, Krukowski K, Huo XJ, Zhou W, Price TJ, Cleeland C, Heijnen CJ. The anti-diabetic drug metformin protects against chemotherapy-induced peripheral neuropathy in a mouse model. PLoS One. 2014 Jun 23;9(6):e100701. doi: 10.1371/journal.pone.0100701. eCollection 2014. PMID 24955774
- [Result] Hershman DL, Lacchetti C, Dworkin RH, Lavoie Smith EM, Bleeker J, Cavaletti G, Chauhan C, Gavin P, Lavino A, Lustberg MB, Paice J, Schneider B, Smith ML, Smith T, Terstriep S, Wagner-Johnston N, Bak K, Loprinzi CL; American Society of Clinical Oncology. Prevention and management of chemotherapy-induced peripheral neuropathy in survivors of adult cancers: American Society of Clinical Oncology clinical practice guideline. J Clin Oncol. 2014 Jun 20;32(18):1941-67. doi: 10.1200/JCO.2013.54.0914. Epub 2014 Apr 14. PMID 24733808
- See also: Pathophysiology of Chemotherapy-Induced Peripheral Neuropathy. — https://www.frontiersin.org/articles/10.3389/fnmol.2017.00174/full